CLINICAL TRIAL: NCT00861367
Title: Prospektive Doppel-Blind-randomisierte Studie Zur Verwendung Von Aspirin Bei Transurethralen Operationen
Brief Title: Prospective Double-blind Study for the Use of Aspirin During Transurethral Surgery of the Bladder or the Prostate
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: difficult enrollment, focus of study no longer of interest
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 05/08
Record Dates: First submitted 2009-03-12; First posted 2009-03-13 (Estimated); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Blood Loss, Surgical; Intraoperative Complications; Re-operation Rates in Patients With Aspirin Treatment
Keywords: aspirin; blood loss; transurethral surgery
MeSH Terms: conditions — Blood Loss, Surgical; Intraoperative Complications; Hemorrhage | interventions — Aspirin

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): aspirin 100mg
  Interventions: Drug: transurethral surgery with or without aspirin
- 2 (Placebo Comparator): empty capsule
  Interventions: Drug: transurethral surgery with or without aspirin

INTERVENTIONS:
Drug: transurethral surgery with or without aspirin — aspirin 100mg once a day, transurethral surgery with or without aspirin
  Other Names: Asprin cardio 100mg

SUMMARY:
Aspirin is very common in older patients. Therefore many of the investigators patients have aspirin. The aim of the study is to proof that Transurethral Surgery of the bladder or the prostate can be performed with aspirin.

ELIGIBILITY:
Inclusion Criteria:

* Transurethral surgery of the bladder or prostate, informed consent, age over 18

Exclusion Criteria:

* Oral anticoagulation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Blood loss | intraoperative, 6 hours post op, 3 days postop

SECONDARY OUTCOMES:
Reoperation rates | during hospitalization

CONTACTS AND LOCATIONS:
Overall Officials: Thomas C Gasser, Prof, Study Chair — Department of Urology, Liestal
Locations (1):
- Urologische Universitätsklinik Basel-Liestal, Liestal, Switzerland